CLINICAL TRIAL: NCT01541319
Title: Mechanism and Repository Study for the Red Cell Storage Duration Study
Acronym: MARS
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 712; 3U01HL072268-09S1 (NIH)
Record Dates: First submitted 2012-02-16; First posted 2012-02-29 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Cardiac Surgery; Erythrocyte Transfusion
Keywords: Cardiac Surgery; Erythrocyte Transfusion

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, pRBCs, PBMCs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Randomized to <= 10day RBCs & transfused: Subjects in the RECESS study who were randomized to receive red blood cell (RBC) units stored no more than 10 days, and who received at least one RBC transfusion between randomization and 96 hours after the cardiac surgery ends
- Randomized to >= 21day RBCs & transfused: Subjects in the RECESS study who were randomized to receive red blood cell (RBC) units stored at least 21 days, and who received at least one RBC transfusion between randomization and 96 hours after the cardiac surgery ends
- Randomized but not transfused: Subjects randomized in the RECESS study who did not receive any red blood cell units between randomization and 96 hours after the end of surgery
- Healthy volunteers

SUMMARY:
A large multicenter randomized controlled trial of approximately 1700 critically ill patients' status post complex cardiac surgery with sternotomy, called the Red Cell Storage Duration Study (RECESS), is currently ongoing. In the RECESS trial, study groups are randomized to either RBCs of less than or equal to 10 days storage time or to greater than or equal to 21 days. The primary outcome of RECESS is a change in multiple organ dysfunction score. Secondary outcomes in RECESS include all cause 28-day mortality, mechanical ventilation free days, and other clinical outcomes. The RECESS study presents a unique opportunity to investigate mechanisms associated with RBC storage duration in the context of clinical outcomes for well-characterized surgical study groups. The ancillary study described here is called the Mechanism and Repository Study (MARS) for RECESS.

The MARS study will analyze the most commonly reported and hypothesized mechanisms considered to be associated with the RBC storage lesion and adverse outcomes in critically ill patients. Laboratories with expertise in RBC function, nitric oxide mechanisms, the coagulation cascade, microparticle analysis and immunology will each examine hypotheses addressing mechanisms potentially able to relate storage time to clinical outcomes in RBC transfusion recipients. At the conclusion of the study, the results will provide a much better understanding of how RBC storage age affects recipient RBC function, coagulation parameters, microparticle load and immune modulation. Perhaps most importantly, this study will also develop a large sample repository for future analysis.

DETAILED DESCRIPTION:
MARS will enroll approximately 250 of the subjects participating in the RECESS study, and an additional 50 healthy volunteers. The RECESS subjects participating in MARS will have blood drawn before their cardiac surgery, and again 2 days after their cardiac surgery. If they have received any red blood cell (RBC) transfusions during their surgery or in the 96 hours following the end of their surgery, they will also have blood drawn at approximately 6 days, 28 days, and 180 days after their surgery, and will answer a health questionnaire at the 28-day and 180-day visits. The healthy volunteers participating in MARS will each have a single blood draw.

All MARS subjects will have blood samples sent to a repository for future study. A subset of the RECESS subjects participating in MARS, and all the healthy volunteers participating in MARS, will also have a number of laboratory tests performed as part of the MARS study. These tests will include

1. laboratory measures of vascular signaling, including NO content, NO disposition; oxidative modification to RBC membrane thiols; and the flux in vasoactive S-nitrosothiols (RSNOs).
2. laboratory measures of coagulation, including thrombin generation; prothrombin fragment 1+2, fibrinopeptide A; soluble thrombomodulin, protein C, PAI-1, tissue plasminogen activator, Factor V, Factor VII, Factor VIII, D-Dimer, antithrombin III, soluble endothelial protein C receptor, TFPI, Xia, INR, PT, and PTT (all using standard testing methods); and clot formation measured by rotation thrombo-elastometry.
3. laboratory measures of microparticle counts, including CD3(T cells), CD66b(Granulocytes), CD 14(Monocytes), CD42a(Platelets), CD235a(RBCs), CD41a(Platelets), CD44(Surface glycoprotein), CD35(Complement receptor1), CD108(Semaphorin 7A), Annexin V, CD154(CD40-ligand), CD62p(p-selectin), CD59(Protectin), CD55(complement DAF), CD58(LFA-3).
4. laboratory measures of inflammation and immune function, including regulatory T cells,Th17 cells, MMP-9, MPO, Pi-1 (total), sE-Selectin, sICAM-1, sVCAM-1, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12 (p70), IL-13, IFN-γ, GM-CSF, and TNF-α.

At one hospital, samples from RBC units transfused to MARS subjects will also be analyzed for nitric oxide parameters.

The primary objective of MARS is to compare post-operative values of these laboratory parameters between RBC-transfused RECESS subjects randomized to receive RBCs stored 10 days or less and RBC-transfused RECESS subjects randomized to receive RBCs stored 21 days or more.

Secondary objectives include

1. Determining whether values of the above laboratory parameters are associated with clinical outcomes among RECESS participants, including change in the multi-organ dysfunction score (MODS) from pre-surgery through death, hospital discharge, or post-operative day 7 (whichever occurs first); change in the MODS from pre-surgery through death, hospital discharge, or post-operative day 28 (whichever occurs first); and all-cause mortality.
2. Determining whether there are correlations between the above laboratory parameters in RECESS subjects at each time point (pre-surgery and post-operative days 2, 6, and 180).
3. Comparing changes in the above laboratory parameters from pre-surgery through Day 2 for randomized RECESS subjects who undergo surgery but do not receive any RBC transfusions versus those in each randomized treatment group who do receive RBC transfusions.
4. Comparing values of the above laboratory parameters in healthy volunteers to pre-surgery values in RECESS subjects scheduled to undergo cardiac surgery.
5. Assessing how nitric oxide parameters in RBC units differ depending on storage duration of the units.
6. Assessing how post-transfusion nitric oxide parameters in transfused subjects differ depending on the pre-transfusion nitric oxide parameters and the parameters in the transfused units.

ELIGIBILITY:
Inclusion Criteria for RECESS subjects participating in MARS:

1. Randomized in Red Cell Storage Duration Study (RECESS)
2. Patients ≥ 18 years old

Exclusion Criteria for RECESS subjects participating in MARS:

* There are no exclusion criteria.

Inclusion Criteria for healthy volunteers participating in MARS:

1. At least 18 years old
2. In generally good health

Exclusion Criteria for healthy volunteers participating in MARS:

1. History of red blood cell transfusion within the previous 6 months.
2. History of surgery within the previous 6 months.
3. Currently treated with inhaled nitric oxide, nitroglycerin in any form, or nitroprusside.
4. Currently treated with prednisone, corticosteroids, cyclosporine, chemotherapy, remicade, methotrexate, Enbrel and/or any antibody based therapy to modulate the immune system.
5. Currently treated with heparin or other anticoagulants (for example coumadin, pradaxa, and low molecular weight heparin).
6. Received any non-steroidal anti-inflammatory drug within the previous 24 hours.
7. Received aspirin within the previous 5 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are two study populations for MARS. One study population is adult subjects undergoing complex cardiac surgery who are participating in the RECESS trial. The other study population is a set of healthy adult volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2012-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Comparison of pre- and post-operative lab values of vascular signaling, coagulation, microparticle counts, and inflammation and immune function | Day 2, 6, 28 and 180
  The primary objective of MARS is to compare post-operative values of these laboratory parameters between RBC-transfused RECESS subjects randomized to receive RBCs stored 10 days or less and RBC-transfused RECESS subjects randomized to receive RBCs stored 21 days or more.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Spinella, MD, Study Chair — Washington University School of Medicine; Philip Norris, MD, Study Chair — Vitalant Research Institute; Susan Assmann, PhD, Principal Investigator — Carelon Research
Locations (13):
- United States (13):
  - Blood Systems Research Institute, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Indiana/Ohio Heart, Fort Wayne, Indiana
  - University of Iowa, Iowa City, Iowa
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - University of Minnesota - Fairview, Minneapolis, Minnesota
  - Robert Wood Johnson Medial School, New Brunswick, New Jersey
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Texas Heart Institute, Houston, Texas
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert Memorial Hospital, Milwaukee, Wisconsin
  - Aspirus Heart & Vascular Institute, Wausau, Wisconsin